CLINICAL TRIAL: NCT05067738
Title: The Development of a Novel Same Day Discharge Program After Pulmonary Resection: A Safety and Feasibility Pilot Study
Brief Title: Same Day Discharge for Wedge Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Rahul Nayak, Director of Research, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: v1.0 7 July 2021
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Surgery; Minor; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 phases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Discharge (Other): Phase 1-Patients will continue to be admitted after their surgery as is the current practice. Phase 2-Patients will have their chest tube removed once they meet chest tube removal criteria and will be discharged home once they meet discharge criteria.
  Interventions: Other: same day discharge

INTERVENTIONS:
Other: same day discharge — same day discharge

SUMMARY:
Monitoring carefully selected participants to determine if participants can be safely discharged the same day of pulmonary resection

DETAILED DESCRIPTION:
Determination of the feasibility of implementing a same day discharge program after minor pulmonary surgery. This will be determined by evaluating the percentage of participants who have chest tubes removed successfully, as well as evaluating the percentage of participants who would be classified as discharged on the day of surgery. The investigators will also be evaluating morbidity associated with this protocol by capturing rates of pleural reintervention.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years of age and older who are scheduled to undergo an elective minimally invasive wedge resection of their lung.

Exclusion Criteria:

1. Pulmonary function tests demonstrating forced expiratory volume in 1 second (FEV1) <50% predicted, FEV1 <1.5L and/or diffusion lung capacity of carbon monoxide (DLCO) <50% predicted.
2. Patient receives an intraoperative pleurodesis.
3. Conversion to open thoracotomy or mini thoracotomy intraoperatively.
4. Active pregnancy.
5. Thoracic Revised Cardiac Risk Index Score (ThRCRI)8 >2.
6. Underlying cognitive disorder resulting in inability to complete activities of daily living.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of successful same day discharge | 2 years
  These patients will have their chest tube removed once they meet chest tube removal criteria and will be discharged home once they meet discharge criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Nayak, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No